CLINICAL TRIAL: NCT03227848
Title: eMurmur ID - Clinical Performance Evaluation
Status: Completed | Type: Observational
Sponsor: CSD Labs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: OTT03
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Heart Murmurs; Pathologic Murmurs; Innocent Murmurs; Congenital Heart Defect; Systolic Murmurs; Diastolic Murmurs
MeSH Terms: conditions — Heart Murmurs; Heart Defects, Congenital; Systolic Murmurs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Automated Heart Murmur Detection AI — Automated AI algorithm-based analysis of digital heart sound recordings to detect and classify heart murmurs. Heart sound recordings were fully blinded before undergoing one-time automated analysis. AI algorithm results for each recording include: AHA classification (Class I (pathologic heart murmur) versus class III (innocent heart murmur or no heart murmur), murmur timing, murmur grade, heart rate and S1/S2 identification.
  Other Names: eMurmur ID

SUMMARY:
The differentiation between innocent and pathologic murmurs through traditional auscultation can often be challenging, which in the end makes the diagnosis strongly dependent on the clinitians experience and clinical expertise. With the development of technology it is now possible to help diagnose heart murmurs using computer aided auscultation systems (CAA). eMurmur ID is an investigational CAA system (not FDA cleared) and the investigators hypothesize that it can distinguish between AHA class I (pathologic murmurs) and AHA class III heart sounds (innocent murmurs and/or no murmurs) with a sensitivity and specificity not worse compared to a similar FDA cleared CAA system on market.

ELIGIBILITY:
Inclusion Criteria:

* All age groups of patients will be included from 1day old
* Patients who are being followed for known congenital heart disease and are returning for follow up
* Patients referred for a suspected heart murmur

Exclusion Criteria:

* Mismatch between the expert physician's diagnosis (auscultation based) and the diagnosis resulting from echocardiography (independently read by a cardiologist blinded to the auscultation results). Note: both, the expert physician and echocardiography results must independently reach the same diagnosis, which is then accepted as the gold standard reference diagnosis to which both devices are compared to. This is necessary because not every pathology visible on an echocardiogram causes an audible murmur, and not every murmur heard by a medical expert might correlate to pathology.
* Patient whose behaviour does not allow for a standard auscultation by the physician (e.g. a screaming fit).

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be chosen based on the heart murmur types required to meet a specified target patient population. Pre-selection of AHA class I and AHA class III patients will be done to achieve a reasonably similar distribution of murmur types compared to a US patient population. All major pathological and innocent murmur types will be included and their occurrence depending on age will be considered. Number of participants drawn: 120 participants across all ages will be included, 75% pediatric and 25% adult.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
eMurmur ID sensitivity and specificity | 1 day
  The primary endpoints of the study are sensitivity and specificity. The clinical reference gold standard diagnosis is defined as expert physicians' diagnosis confirmed by independently interpreted echocardiogram diagnosis.
  True positive (TP), true negative (TN), false positive (FP) and false negative (FN) will be determined via comparison of the heart murmur classification results with the clinical gold standard (echocardiogram) diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Lai, MD, Principal Investigator — Children's Hopsital of Eastern Ontario, Canada
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai LS, Redington AN, Reinisch AJ, Unterberger MJ, Schriefl AJ. Computerized Automatic Diagnosis of Innocent and Pathologic Murmurs in Pediatrics: A Pilot Study. Congenit Heart Dis. 2016 Sep;11(5):386-395. doi: 10.1111/chd.12328. Epub 2016 Mar 15. PMID 26990211
- See also: Computerized Automatic Diagnosis of Innocent and Pathologic Murmurs in Pediatrics: A Pilot Study. — https://www.ncbi.nlm.nih.gov/pubmed/26990211